CLINICAL TRIAL: NCT01364662
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of SPN-810 as Adjunctive Therapy in Children With Impulsive Aggression Comorbid With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A Study to Evaluate the Efficacy and Safety of SPN-810 as Adjunctive Therapy in Children With Impulsive Aggression Comorbid With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 810P202
Record Dates: First submitted 2011-05-25; First posted 2011-06-02 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2015-11

CONDITIONS: Impulsive Aggression Comorbid With ADHD
Keywords: Impulsive Aggression; Attention Deficit Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: SPN-810
- 3 (Experimental)
  Interventions: Drug: SPN-810
- 4 (Experimental)
  Interventions: Drug: SPN-810

INTERVENTIONS:
Drug: SPN-810 — administered orally
  Arms: 2; 3; 4
Drug: Placebo — administered orally
  Arms: 1

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, dose-ranging, efficacy and safety study in children with impulsive aggression comorbid with Attention-Deficit/Hyperactivity Disorder (ADHD). The target subjects are healthy male and female children aged 6 to 12 years, inclusive, with a diagnosis of ADHD. A total of 120 subjects will be randomized across approximately 30 US centers to one of four treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pediatric male or female subjects, age 6 to 12 years.
2. Diagnostic and Statistical Manual of Mental Disorders - IV -Text Revision (DSM-IV-TR) diagnosis of ADHD.
3. R-MOAS score >=24 at screening and R-MOAS score >=20 for randomization
4. IQ greater than 71.
5. Weight of >=20kg
6. current treatment with psychostimulant (1 month prior to screening)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Reduction in aggressive behavior as assessed by R-MOAS score | Change from baseline to Visit 10

SECONDARY OUTCOMES:
Safety of SPN-810 Safety as assessed by safety scales, AEs, clinical labs, vitals, Physical Exams, and ECGs | Visit 2 to End of Study
  Safety as assessed by safety scales, AEs, clinical labs, vitals, Physical Exams, and ECGs
Change in CGI-S | Baseline to Visit 5
CGI-I score at each post-baseline Visit | Baseline to Visit 5
Change in SNAP-IV ADHD scores | Baseline to Visit 5

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Dothan, Alabama
  - Los Angeles, California
  - Santa Ana, California
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Maitland, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Libertyville, Illinois
  - Indianapolis, Indiana
  - Terre Haute, Indiana
  - Owensboro, Kentucky
  - Toms River, New Jersey
  - Stony Brook, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Bellevue, Washington
  - Bothell, Washington